CLINICAL TRIAL: NCT04225130
Title: Decreasing Suicide Risk Among Service Members With Posttraumatic Stress Using Written Exposure Therapy
Brief Title: Decreasing Suicide Risk Among Service Members With Posttraumatic Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston VA Research Institute, Inc. (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Brian Marx, PH.D., Deputy Director, Behavioral Science Division, National Center for PTSD, Boston VA Research Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W81XWH-16-2-0003
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Suicide; Posttraumatic Stress Disorder
MeSH Terms: conditions — Suicide; Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written Exposure Therapy -for Suicide (Experimental): Written Exposure Therapy-for Suicide (WET-S) consists of 5 treatment sessions. Each session includes a written exposure exercise. It also includes CRP. Participants assigned to WET-S will complete the CRP prior to beginning their writing in session 1. Patient use of the CRP since the previous session will be briefly reviewed at the start of each WET-S session to manage safety and problem solve fluctuations in risk during treatment.
  Interventions: Behavioral: Written Exposure Therapy -for Suicide
- Treatment as Usual (Active Comparator): The TAU condition consists of daily contact and patient centered care by the acute psychiatric inpatient unit provider team. TAU includes initial stabilization, nurse case management, medication management, psychoeducation groups, and discharge planning. Patients engage with the provider team daily.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Written Exposure Therapy -for Suicide — The first session will consist of the therapist educating the participant about common reactions to trauma and providing information regarding the rationale of WET-S as a treatment for PTSD. The participant will then be given general instructions for completing the trauma narratives, specific instructions for completing the first session, and will then complete the first (30 minutes) narrative writing session. Participants will be instructed to write about the same trauma experience during each session. The importance of delving into their deepest emotions surrounding the trauma event is emphasized. All WET-S sessions will take place in a private room and begin with the therapist reading the specific writing instructions for that session and then leaving the instructions with the participant while 30-minute writing session is completed.
  Other Names: WET-S
  Arms: Written Exposure Therapy -for Suicide
Behavioral: Treatment as Usual — The TAU condition consists of daily contact and patient centered care by the acute psychiatric inpatient unit provider team (e.g., psychiatrists, therapists, case managers, behavioral health techs). TAU includes initial stabilization, nurse case management, medication management, psychoeducation groups, and discharge planning. Patients engage with the provider team daily.
  Other Names: TAU
  Arms: Treatment as Usual

SUMMARY:
In this study, the investigators will conduct a randomized controlled trial (RCT) to evaluate the efficacy of the WET-S + treatment as usual (TAU) compared with TAU among high-risk, suicidal service members with PTSD or posttraumatic stress (PTS) admitted to the Carl R. Darnall Army Medical Center (CRDAMC) acute inpatient psychiatry unit at Fort Hood, Texas. Suicide risk and PTS symptom severity are the primary outcomes. Secondary outcomes include subsequent hospitalizations for suicidal thoughts and behaviors and suicide attempts. Investigators will conduct a needs assessment with stakeholders during the RCT to develop a tool kit for WET implementation in other DoD inpatient psychiatry units.

DETAILED DESCRIPTION:
This study aims to compare a new formulation of WET referred to as WET-for suicide (WET-S) that includes crisis response planning + treatment as usual (TAU) compared with TAU among high-risk, suicidal service members with PTS admitted to the Carl R. Darnall Army Medical Center (CRDAMC) acute inpatient psychiatry unit at Fort Hood, Texas.

Aim 1: Determine if WET-S reduces the presence, frequency, and severity of suicidal ideation, suicide plans, suicide gestures, suicide attempts, non-suicidal self-injurious behaviors, and rehospitalization for suicidality.

Aim 2: Determine if WET-S + TAU reduces PTS symptom severity among service members admitted to an acute psychiatric inpatient unit for SI and/or attempt compared with TAU.

Aim 3: Determine if reductions in PTS symptoms mediate the association between treatment condition and suicide-related outcomes (suicidal ideation, plans, gestures, attempts, non-suicidal self-injurious behaviors, and rehospitalizations).

Aim 4: Develop a tool kit for WET-S implementation through a needs assessment with key stakeholders and evaluation of contextual factors among DoD inpatient facilities to determine readiness for successful implementation of WET-S.

Study investigators will conduct a randomized controlled trial (RCT) to evaluate the efficacy of the WET-S + treatment as usual (TAU) compared with TAU among high-risk, suicidal service members with PTSD or posttraumatic stress (PTS) admitted to the Carl R. Darnall Army Medical Center (CRDAMC) acute inpatient psychiatry unit at Fort Hood, Texas. Investigators will conduct a needs assessment with stakeholders during the RCT to develop a tool kit for WET implementation in other DoD inpatient psychiatry units.

Data will be collected in Texas. Investigators conservatively anticipate enrollment of approximately 140 service members to achieve a final sample size of 124 (n = 62 per condition) after accounting for 15% attrition. CRDAMC receives approximately 4500 admissions each year for SI/attempt. TAU on the inpatient unit consists of crisis management and stabilization. Suicide risk and PTS symptom severity are the primary outcomes. Secondary outcomes include subsequent hospitalizations for suicidal thoughts and behaviors and suicide attempts.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older) service members hospitalized at Carl R Darnall Army Medical Center for SI/suicide plan or attempt.
* Symptoms of posttraumatic stress (PTS) of at least moderate severity (total scores > 20) confirmed by assessor using the CAPS-5.
* Speak, read, and write English.

Exclusion Criteria:

* Active psychosis.
* The presence of moderate to severe cognitive impairment (as determined by the inability to comprehend the baseline screening questionnaires).
* The presence of any factor that may impair an individual's ability to comprehend and effectively participate in the study, including the presence of extreme agitation or violent behavior.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Clinician Administered PTSD Scale Scores | baseline, 1-month, 4-month follow-up
  The CAPS-5 is a structured diagnostic interview and gold standard for assessing PTSD. It provides a dichotomous PTSD diagnosis and overall symptom severity score. Scores range from 0 to 80, with greater scores signifying more severe PTSD symptoms.
Change in Self-Injurious Thoughts and Behaviors Interview Scores | Baseline, 1-month, 4-month follow-up
  The SITBI is a structured interview that assesses the presence (lifetime, past year, past month), frequency, severity, and characteristics of five types of SITB: (a) suicidal ideation, (b) suicide plans, (c) suicide gestures, (d) suicide attempts, and (e) non-suicidal self-injury. The SITBI assesses the frequency of each type of thought or behavior in the respondent's lifetime, past year, and past month, as well as the age of onset of each thought or behavior endorsed. The SITBI also assesses the severity of each thought or behavior endorsed on a scale from 0 (low/little) to 4 (very much/severe) scale, on average and at the worst point at each of those time frames.
Change in medical record outcomes | Baseline, 1-month, 4-month follow-up
  At baseline and each follow-up assessment, study staff will access participants' medical record to obtain information about current and past mental health treatment, current and past psychiatric diagnoses, current and past psychiatric medication, and history of suicidal thoughts and behaviors. If applicable, date of admission(s) to inpatient psychiatric unit, chief complaint at the time of admission(s), details of psychiatric stay(s), and length of stay(s) will also be obtained. Changes in any of these variables from baseline to follow-up will be recorded.
Change physical and mental health assessed by Military Suicide Research Consortium Common Data Elements | Baseline, 1-month, 4-month follow-up
  Participants will provide self-report information about their physical and mental health and behaviors at each time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Carl R Darnell Army Medical Center, Fort Hood, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from study participants will be prepared and stored in the Military Suicide Research Consortium data repository, where it can then be accessed by interested researchers.
Time Frame: Per the agreement with MSRC, the data will be placed in the repository periodically. Following completion of the study and publication of papers focused on primary study aims, the data will be available. There is no time limit for how long it will be available.

REFERENCES:
- [Derived] Kearns JC, Straud CL, Stanley IH, Sloan DM, Fina BA, Young-McCaughan S, Tyler HC, Kaplan AM, Blankenship AE, Schrader CC, Green VR, Bryan CJ, Peterson AL, Marx BP; STRONG STAR Consortium. Written Exposure Therapy for Posttraumatic Stress Symptoms and Suicide Risk: A Randomized Controlled Trial With High-Risk Patients Admitted to a Military Inpatient Psychiatric Unit. Suicide Life Threat Behav. 2025 Apr;55(2):e70008. doi: 10.1111/sltb.70008. PMID 40052305

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT04225130/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT04225130/ICF_001.pdf